CLINICAL TRIAL: NCT04972331
Title: Arthroscopic Partial Menisectomy or Platelet Rich Plasma in Degenerative Meniscus Without Osteoarthritis? Study Protocol for a Randomized Controlled Trial
Brief Title: Degenerative Meniscus Without Osteoarthritis : Arthroscopic Partial Menisectomy Versus Platelet Rich Plasma (APM-PRP)
Acronym: APM-PRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Chirurgie Reparatrice Locomoteur et Sports (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-090107-01
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Meniscectomy; Platelet-Rich Plasma; Meniscus; Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Active Comparator): Arthroscopic Partial menisectomy
  Interventions: Procedure: Arthroscopic Partial Meniscectomy; Other: Post-intervention
- INTERVENTION (Experimental): Platet- Rich-Plasma
  Interventions: Procedure: Platet- Rich-Plasma; Other: Post-intervention

INTERVENTIONS:
Procedure: Arthroscopic Partial Meniscectomy — Arthroscopic partial meniscectomy was performed by three senior surgeons using two standard portals, no outflow cannula, a 5.5-mm 30° arthroscope, and a pressure-controlled irrigation system.
  A standard surgical protocol was used to document possible findings in the cartilage, ligaments, synovium, and medial and lateral meniscus. In each case, surgery was limited to resection with limited debridement of the articular surface lesion, preserving as much of the meniscus as possible. Patients who underwent additional procedures, such as removal of loose bodies or subchondral drilling for any articular lesions, were excluded from this study (Figure 1). No patients underwent total meniscectomy or meniscal repair.
  Arms: CONTROL
Procedure: Platet- Rich-Plasma — Peripheral venous blood was collected from all patients, which was then centrifuged to isolate red blood cells from the upper plasma layer. We used the Arthrex® kit APC®. The upper plasma layer was carefully collected with a serological pipette and placed in a new centrifuge tube or set aside for injection. The 5 mL remaining upper plasma layer was centrifuged again to separate platelet-poor plasma from PRP for 7 min. We activated the PRP sample by adding calcium chloride through ultraviolet irradiation, and then a 4- to 8-mL sample was used for two injections. One injection was performed intra-articularly with a supero-lateral approach. One ultrasound-guided injection was performed at the meniscal wall. Our protocol allowed us to have < 1% blood cells and <1% white cells in the injection.
  Arms: INTERVENTION
Other: Post-intervention — All patients were discharged the day after surgery with no limitation of mobility but with restrictions on sports for four weeks. Interruption of work was given for 10-45 days. The same analgesics and NSAIDs were administered in both groups for two weeks. All patients then received a rehabilitation program conducted by a physiotherapist, using the same protocol as in the PRP group for four weeks.

SUMMARY:
This study compares arthroscopic partial menisectomy (APM) and platelet rich plasma (PRP) for degenerative meniscal injury of the knee.

The current state of knowledge is poor. There are few comparative studies that have been performed and only on surgical treatment or rehabilitation. Moreover, these studies show contradictory results.

The main objective of this study is to compare APM and PRPinfiltration, in terms of pain reduction, which is greater with the surgical technique than in the PRP infiltration group.

The hypothesis of this study is that there is superiority of surgery over PRP infiltration.

The main evaluation criterion is the pre-post-operative pain by a simplified numerical scale.

DETAILED DESCRIPTION:
Degenerative meniscal tear is a chronic, slowly evolving condition that typically involves horizontal cleavage of the meniscus and affects middle-aged men and women. The prevalence is high, with a medial meniscal tear found on imaging in 13-28% of persons older than 50 years of age. In the absence of evidence of knee osteoarthritis, only 22% of patients with meniscal tears have knee symptoms. Symptomatology is internal knee pain, often related to activities or positions such as squatting or kneeling, and usually improves with rest. The optimal treatment for nontraumatic degenerative meniscal tears is currently controversial.

Arthroscopic partial meniscectomy (APM) is one of the most commonly performed orthopedic surgical procedures for patients with meniscal degeneration to improve knee function and reduce pain. However, there is no reliable evidence that arthroscopic partial meniscectomy improves outcomes in the middle-aged population with degenerative meniscal disease. A study comparing APM with sham surgery found no significant difference for APM at six months and at one year with a slightly better outcome for APM at two months. A meta-analysis showed that APM combined with medical exercise leads to a better outcome than isolated medical exercise in immediate follow-up at two months, but there is no difference at 6 months.

Thorlund et al. reported that the effect of knee arthroscopy for degenerative knee (meniscal tears with or without osteoarthritis) was limited at 3-6 months after the procedure with 0.17 to 0.96% venous embolism.

A recent study reported a 15.7% conversion rate from APM to Total Knee Arthroplasty (TKA) at 10 years postoperatively.

There are numerous types of infiltrations with the goal of a pain-free knee. Hyaluronic acid (HA), might have a healing-promoting effect and tend to delay the need for APM, but this effect is still controversial and has not been verified in studies. There is increasing clinical interest in testing new biological products to improve the efficacy of intra-articular injection treatment.

Platelet-rich plasma (PRP) is an autologous whole blood extract containing high concentrations of platelets and growth factors that promises to promote and accelerate recovery of injured ligaments, muscles, tendons, and joints by injecting the patient's own platelets. It has few side effects and can be performed in a consultation setting. It is still controversial and results are inconsistent, which could be due to the use of leukocyte-poor PRP or leukocyte-rich PRP, which have different functions such as anti-infectious actions and immune regulation. Moreover, there is confusion between PRP and platelet-rich fibrin (PRF).

Regarding knee osteoarthritis and the comparison with HA, 11 meta-analyzes came to positive conclusions and 2 contradicted the efficacy.

Regarding injection of PRP into a degenerative meniscal lesion, functional outcomes appear to improve and failure rates decrease. In a case-control study of open meniscal repair of horizontal tears in young patients, the addition of PRP slightly improved clinical outcomes at mid-term follow-up.

Nonoperative treatment has a conversion rate to surgery in 0 to 35% of patients. Meanwhile, osteoarthritis after meniscectomy is common. In a multicenter study from French Arthroscopy Society, the prevalence of joint line narrowing in the medial meniscus was 22% with a mean follow-up of 13 years.

There are several treatment options for symptomatic degenerative meniscal tears. However, to the investigators' knowledge, there is no report on PRP and no results comparing APM and PRP have been reported.

Therefore, the aim of this study is to compare two treatments; APM and PRP, both followed by rehabilitation, in terms of knee pain, knee function and satisfaction in patients with degenerative meniscal tears without osteoarthritis. The hypothesis is that APM would be superior than PRP in terms of pain and functional outcomes at 3 months postoperative

ELIGIBILITY:
Inclusion Criteria:

* Eligible for APM
* Acceptance of infiltration procedure or APM
* Patient age above 30 years and under 65 years
* Acceptance of outpatient procedure
* Non-locked painful knee ≥ 1 month
* No osteoarthritis Kellgren-Lawrence ≤ 2 or Alhback ≤ 1 (Monopodal weh-ight-bearing AP and profile X-Ray with the knee in extension and bipedal schuss X-Ray with the knee at 45° of flexion
* No malignment > 5° (Full leg standing X-Ray)
* Pain when squatting
* Medial pain
* MRI confirmed unique horizontal degenerative medial lesion

Exclusion Criteria:

* Traumatic meniscal injury
* Neurological or rheumatic inflammatory diseases
* MRI : Loose bodies or ligament injuries or osteochondral defects or tumors
* Previous ipsilateral knee surgery

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 3 months
  Scale from 0 to 10 to evaluate pain (0 is no pain and 10 is worse pain ever)

SECONDARY OUTCOMES:
Simple Knee Value (SKV) | Preop, 1 month, 2 months, 3 months, 6 months, 12 months
  Scale from 0 to 100 to evaluate the knee function in daily life (0 is no function and 100 is normal function)
Knee injury and Osteoarthritis Outcome Score (KOOS) | Preop, 1 month, 2 months, 3 months, 6 months, 12 months
  To assess the patient's opinion about their knee and associated problems from 0 worse function to 152 best function, also reported to % by dividing by 152
IKDC score (from International Knee Documentation Committee) | Preop, 1 month, 2 months, 3 months, 6 months, 12 months
  Subjective evaluation of the knee function (from 0 to 100%, 0 is no function and 100 is normal function)
Lysholm Score | Preop, 3 months, 6 months, 12 months
  Activity of the knee after injuries (scale from 0 to 100 where 0 is no activity and 100 is normal activities
Net Promoter Score (NPS) | 3 months, 6 months, 12 months
  whether or not the patient recommended the questionnaire used, a scale of 0 (not at all likely) to 10 (very likely)
Healing meniscus | 6 months
  Healing meniscus on MRI (normal signal intensity of tear on T2-weighted imaging is consider as healed, intermediate, bright, or fluid is not healed)
Osteoarthritis grade (Alhback classification) | 3 months, 6 months, 12 months
  Progression of osteoarthritis on X-rays with Alhback classification

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Boileau, MD,PhD, Study Chair — ICR-Nice
Locations (1):
- ICR Clinique Kantys Centre, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aprato A, Sordo L, Costantino A, Sabatini L, Barberis L, Testa D, Masse A. Outcomes at 20 Years After Meniscectomy in Patients Aged 50 to 70 Years. Arthroscopy. 2021 May;37(5):1547-1553. doi: 10.1016/j.arthro.2020.11.053. Epub 2020 Dec 9. PMID 33307147
- [Background] Braun HJ, Wasterlain AS, Dragoo JL. The use of PRP in ligament and meniscal healing. Sports Med Arthrosc Rev. 2013 Dec;21(4):206-12. doi: 10.1097/JSA.0000000000000005. PMID 24212368
- [Background] Vermesan D, Prejbeanu R, Laitin S, Damian G, Deleanu B, Abbinante A, Flace P, Cagiano R. Arthroscopic debridement compared to intra-articular steroids in treating degenerative medial meniscal tears. Eur Rev Med Pharmacol Sci. 2013 Dec;17(23):3192-6. PMID 24338461
- [Background] Yim JH, Seon JK, Song EK, Choi JI, Kim MC, Lee KB, Seo HY. A comparative study of meniscectomy and nonoperative treatment for degenerative horizontal tears of the medial meniscus. Am J Sports Med. 2013 Jul;41(7):1565-70. doi: 10.1177/0363546513488518. Epub 2013 May 23. PMID 23703915
- [Background] Thorlund JB, Hare KB, Lohmander LS. Large increase in arthroscopic meniscus surgery in the middle-aged and older population in Denmark from 2000 to 2011. Acta Orthop. 2014 Jun;85(3):287-92. doi: 10.3109/17453674.2014.919558. Epub 2014 May 6. PMID 24800623